CLINICAL TRIAL: NCT02029456
Title: Low Dose Prolonged Infusion of Tissue Type Plasminogen Activator Therapy in Massive Pulmonary Embolism: AYKAN Trial
Brief Title: Low Dose Prolonged Infusion of Tissue Type Plasminogen Activator Therapy in Massive Pulmonary Embolism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, AHMET CAGRI AYKAN, Medical Doctor,, Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 538.38792-903/6190
Record Dates: First submitted 2013-11-17; First posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Pulmonary Embolism
Keywords: Massive Pulmonary embolism; thrombolytic therapy; high risk; elderly
MeSH Terms: conditions — Pulmonary Embolism | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low dose prolonged infusion arm (Experimental): Low dose prolonged infusion of tPA arm (25mg Actilyse in 6 hours)
  Interventions: Drug: 25 mg Actilyse ( Boehringer Ingelheim, Germany) infusion in 6 hours

INTERVENTIONS:
Drug: 25 mg Actilyse ( Boehringer Ingelheim, Germany) infusion in 6 hours

SUMMARY:
The aim of the present study was to assess the effects of low-dose (25mg) prolonged administration (in 6 hours) of tissue type plasminogen activator (tPA) on in-hospital mortality and outcomes in patients with massive PE.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is life threatening disease requiring early diagnosis and treatment. Thrombolytic therapy (TT) is required in patients with massive PE. PE has a high mortality but the in-hospital all-cause case mortality rates were lower in unstable patients who received TT than those who did not. However, it was reported that minority (nearly 30%) of unstable patients received thrombolytic therapy. The reason that majority of unstable patients failed to receive thrombolytic therapy is unclear. The higher rates of complications including the life threatening bleeding may be a reason of reluctance in the use of TT.

The lungs are the only organ receiving the entire cardiac output. Therefore, they are the point of convergence for the entire molecules of the thrombolytic agent, independent from the route of administration. So that lower doses of the TT might be effective in PE, with the additional benefits of enhancing its safety profile. The percutaneous endovenous intervention for deep venous thrombosis has suggested an exquisitely favorable pulmonary response to low-dose thrombolysis. The aim of the present study was to assess the effects of low-dose (25mg) prolonged administration (in 6 hours) of tissue type plasminogen activator (tPA) on in-hospital mortality and outcomes in patients with massive PE.

The primary end points consisted of in hospital all cause mortality, major complications, pulmonary hypertension and right ventricular dysfunction. Secondary points are all cause mortality, pulmonary hypertension and right ventricular dysfunction at 6 month.

ELIGIBILITY:
Inclusion Criteria:

Patients with massive PE aged 18 years or older with confirmed PE and able to give informed consent will be included in the study. PE is defined according to current guidelines as adult patients presenting with signs and symptoms suggestive of PE plus imaging documentation on computed tomography angiography. Massive PE was defined as acute PE with sustained hypotension (systolic blood pressure<90 mm Hg for at least 15 minutes or requiring inotropic support, not due to a cause other than PE, such as arrhythmia, hypovolemia, sepsis, or left ventricular [LV] dysfunction), pulselessness, or persistent profound bradycardia (heart rate<40 bpm with signs or symptoms of shock).

Exclusion Criteria:

Patients with prior intracranial hemorrhage, known structural intracranial cerebrovascular disease (eg, arteriovenous malformation), known malignant intracranial neoplasm, ischemic stroke within 3 months, suspected aortic dissection, active bleeding or bleeding diathesis, recent surgery encroaching on the spinal canal or brain, and recent significant closed-head or facial trauma with radiographic evidence of bony fracture or brain injury were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-03 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
All cause in hospital mortality | participants will be followed for the duration of hospital stay, an expected average of 7 days
  Death occured during hospitalization period.
Major complications | participants will be followed for the duration of hospital stay, an expected average of 7 days.
  Major bleeding, intracranial bleeding, resuscitated cardiac arrest, thromboembolism and stroke are described as major complications.
Development of pulmonary hypertension | participants will be followed for the duration of hospital stay, an expected average of 7 days
  Pulmonary artery systolic pressure >40mmHg measured by transthoracic echocardiography prior to discharge was described as pulmonary hypertension.
Right Ventricular dysfunction | participants will be followed for the duration of hospital stay, an expected average of 7 days
  Right ventricular dysfunction detected by transthoracic echocardiography:
  1. Decreased right ventricular diameter (at least 25% decrease of Right ventricle/Left ventricle diameter)
  2. Tricuspid annular plane systolic excursion>16mm)
  3. s'> 10.0 cm/s
  4. Tissue Doppler derived right ventricle myocardial performance index>0.55
Restoration of hemodynamic status | 6 hours after the beginning of thrombolytic therapy
  Systolic blood pressure >100mmHG

SECONDARY OUTCOMES:
Pulmonary hypertension | 6 month
  Pulmonary artery systolic pressure >40mmHg
Right ventricular dysfunction | 6 months
  1. Tricuspid annular plane systolic excursion >16mm
  2. s'> 10.0 cm/s
  3. Tissue Doppler derived right ventricle myocardial performance index>0.55
  4. Right ventricle/Left ventricle diameter <1

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Ç AYKAN, MD, Study Chair — Department of Cardiology, Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital
Locations (1):
- Department of Cardiology, Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital, Trabzon, Turkey (Türkiye)

REFERENCES:
- [Result] Ozkan M, Cakal B, Karakoyun S, Gursoy OM, Cevik C, Kalcik M, Oguz AE, Gunduz S, Astarcioglu MA, Aykan AC, Bayram Z, Biteker M, Kaynak E, Kahveci G, Duran NE, Yildiz M. Thrombolytic therapy for the treatment of prosthetic heart valve thrombosis in pregnancy with low-dose, slow infusion of tissue-type plasminogen activator. Circulation. 2013 Jul 30;128(5):532-40. doi: 10.1161/CIRCULATIONAHA.113.001145. Epub 2013 Jun 28. PMID 23812180
- [Result] Ozkan M, Gunduz S, Biteker M, Astarcioglu MA, Cevik C, Kaynak E, Yildiz M, Oguz E, Aykan AC, Erturk E, Karavelioglu Y, Gokdeniz T, Kaya H, Gursoy OM, Cakal B, Karakoyun S, Duran N, Ozdemir N. Comparison of different TEE-guided thrombolytic regimens for prosthetic valve thrombosis: the TROIA trial. JACC Cardiovasc Imaging. 2013 Feb;6(2):206-16. doi: 10.1016/j.jcmg.2012.10.016. PMID 23489534